CLINICAL TRIAL: NCT04477447
Title: Multicenter PMCF Study on the Safety and Performance of CESPACE 3D - A Prospective Study on Total Indications
Brief Title: PMCF Study on the Safety and Performance of CESPACE 3D
Acronym: CATALINA
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2004
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Degenerative Instability; Spondylolisthesis; Post-discectomy Syndrome; Post-traumatic Instabilities
Keywords: Cervical Vertebrae;; Spondylolisthesis;; Treatment Outcome;; Interbody Fusion
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Prospective, pure data collection of all CeSPACE 3D patients in selected centers (not interventional, multicenter)

ELIGIBILITY:
Inclusion Criteria:

* Patient is minimum 18 years old
* Written informed consent for the documentation of clinical and radiological results
* Patient's indication according to IFU
* Patient is not pregnant

Exclusion Criteria:

• Patient is not willing or able to participate at the follow-up examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Change of Neck Specific Disability measured by Neck Disability Index (NDI) | preoperative, 12 months postoperative
  The NDI is designed to measure neck-specific disability. The questionnaire has 10 items to measure patient-reported disability secondary to neck pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation and patients rate their status from 0 (best) to 5 (worst imaginable). Individual item responses are summed to a total score, where 0 points indicate no activity limitations and 50 points indicate complete activity limitation.

SECONDARY OUTCOMES:
JOA score | preoperatively and at one follow-up- assessment after a minimum of one year postoperatively
  The Japanese Orthopaedic Association (JOA) score is a widely used tool to assess the severity of clinical symptoms in patients with cervical compressive myelopathy. Motor function (Upper extremity/Lower extremity); Sensory (Upper extremity/lower extremity/trunk); Bladder function. The Score reaches a maximum of 17 and a Minimum of 0 points.
Pain (VAS) | preoperatively and at one follow-up- assessment after a minimum of one year postoperatively
  The visual analogue scale (VAS) is a scale used to determine the pain intensity experienced by individuals. It consists of a line, approximately 10-15 cm in length, with the left side signifying no pain with a smiling face image and the right side signifying the worst pain ever with a frowning face image.
development of EQ-5D-5L | preoperatively and at one follow-up- assessment after a minimum of one year postoperatively
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
development of radiological outcome | preoperatively and at one follow-up- assessment after a minimum of one year postoperatively
  if provided in the clinical standard; e.g. fusion, implant subsidence, implant migration)
Rate of AE/SAEs | preoperatively, intraoperatively and at one follow-up- assessment after a minimum of one year postoperatively
  Rate of AE/SAEs during the postoperative course
Patient Satisfaction with Treatment Outcome | at one follow-up- assessment after a minimum of one year postoperatively
  Patient satisfaction with Outcome of surgery documented in two aspects: is the Patient satisfied (four Point scale: very satisfied, satisfied, unsatisfied, very unsatisfied) and would the Patient like to undergo surgery again (yes, no, not willing to say)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Nikolaus Kroppenstedt, Dr. med., Principal Investigator — Abteilung für Wirbelsäulenchirurgie Sana Kliniken Sommerfeld; Francis Kilian, Dr. med., Principal Investigator — Katholisches Klinikum Koblenz
Locations (2):
- Germany (2):
  - Katholisches Klinikum Koblenz, Koblenz
  - Sana Kliniken Sommerfeld, Kremmen